CLINICAL TRIAL: NCT00721617
Title: Free Fatty Acids-Induced Hypertension, Endothelial Dysfunction, Inflammation, Insulin Resistance, and Autonomic Dysfunction in Lean and Obese Subjects
Brief Title: FFA Hypertension and Inflammation in Lean and Obese Subjects
Acronym: FFAADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00009277
Record Dates: First submitted 2008-06-26; First posted 2008-07-24 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes; Hypertension; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Obesity | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obese subjects (Active Comparator): Obese normotensive subjects will receive 24 hour challenges on 3 separate occasions, in a random order, with IV Normal Saline at 20ml/hour, IV Intralipid (20% solution at 20 ml/hour and an oral fat load (96g/24 hours)
  Interventions: Other: Intralipid 20%; Other: Normal Saline; Other: Oral fat load
- Lean subjects (Active Comparator): Lean normotensive subjects will receive 24 hour challenges on 3 separate occasions, in a random order, with IV Normal Saline at 20ml/hour, IV Intralipid (20% solution at 20 ml/hour and an oral fat load (96g/24 hours)
  Interventions: Other: Intralipid 20%; Other: Normal Saline; Other: Oral fat load

INTERVENTIONS:
Other: Intralipid 20% — Lean and obese normotensive subjects will receive Intralipid 20% infusion. Intralipid is an oil-in-water emulsion derived from egg phospholipids, soybean, and glycerol. The Intralipid 20% long-chain triglyceride emulsion contains: 200 g of soy bean oil; 12 g of egg yolk; 25 g of glycerol. The emulsion is composed of the following free fatty acids (FFAs): linoleic acid: 50%, oleic acid: 26%, palmitic acid: 10%, stearic acid: 9%, egg yolk, phospholipids: 3.5% It will be given intravenously at 20 ml/hr (96 g/24 h) for 24 hours.
Other: Normal Saline — Lean and obese normotensive subjects will receive normal saline at 20 ml/hr for 24 hours.
Other: Oral fat load — Lean and obese normotensive subjects will receive an oral fat load at 96 g/24hr. The oral liquid fat load will be given in equal amounts (16 g) every 4 hours (total 96 g over 24 hours).

SUMMARY:
Although a large number of obese patients develop high blood pressure, the cause is unknown. The purpose of this study is to look at the effect of high fatty acids (a type of fat) in the development of high blood pressure in obese people.

DETAILED DESCRIPTION:
Recent studies indicate that increased levels of a circulating fat (free fatty acids or FFAs) increases blood pressure, impairs endothelial (vascular) function, and increases inflammatory markers in subjects with and without diabetes. The effects of FFA on blood pressure and vasculature have not been fully investigated. A group of 12 obese nondiabetic, normotensive subjects will be admitted to the Grady Clinical Research Center (GCRC) on separate 4 occasions. Research subjects will receive, in random order, a 8-hour intravenous (IV) infusion of Intralipid 20% at 40 mL/h (a fat solution), 8-hour IV infusion of normal saline at 40 mL/h, 8-hour IV infusion of dextrose (sugar) 10% at 40 mL/h, and a 8-hour intravenous (IV) infusion combination of Intralipid 20% and dextrose 10% at 40mL/h.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Obese subjects (body mass index (BMI) ≥ 30 kg/m^2)
* 18 and 65 years
* Blood pressure reading < 140/80 mm Hg and no prior history of hypertension

Exclusion Criteria:

* History of diabetes mellitus
* History of hypertension
* Fasting triglyceride levels > 250 mg/dL
* Liver disease (ALT 2.5x > upper limit of normal)
* Serum creatinine ≥1.5 mg/dL
* Smokers, drug or alcohol abuse
* Mental condition rendering the subject unable to understand the scope and possible consequences of the study
* Female subjects who are pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Grady Memorial Hospital
Pre-assignment Details: All subjects had a 2-hour glucose of less than 200 mg/dL during a 75 g oral glucose tolerance test and a fasting glucose of less than 126 mg/dL.
Groups:
- Healthy Subjects: Obese, normotensive, healthy subjects received, in a random order, on four separate occasions, Intralipid 20% at 40 mL/h, dextrose 10% at 40mL/h, combination intralipid 20% and dextrose 10% at 40 mL/h, or normal saline at 40 mL/h
Period: 0 Hour (Baseline) of Saline Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Saline Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 8 Hours Into Saline Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 0 Hour (Baseline) of Intralipid Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Intralipid Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 8 Hours Into Intralipid Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 0 Hour (Baseline) of Dextrose Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Dextrose Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 8 Hours Into Dextrose Infusion
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 0 Hour (Baseline) of Intralipid/Dextrose
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 4 Hours Into Intralipid/Dextrose
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0
Period: 8 Hours Into Intralipid/Dextrose
Arm/Group | Healthy Subjects
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation From Baseline to 4 Hours
Description: Endothelium-dependent brachial artery flow-mediated dilation (FMD) was assessed. Ultrasound images of the brachial artery were obtained and arterial diameters were measured with customized software. FMD is expressed as the change in diameter from baseline to 4 hours.
Time Frame: Baseline, 4 hours
Measure: Mean (Standard Deviation); unit: percent change in diameter
Groups:
- Healthy Subjects: Subjects received either IV Normal Saline at 20ml/hour, IV Intralipid (20% solution at 20 ml/hour and an oral fat load (96g/24 hours) in a random order.
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
percent change in diameter
  Saline | 0.16 (4.9)
  Intralipid 20% | -3.2 (1.4)
  Dextrose 10% | -0.9 (1.8)
  Intralipid/Dextrose | -2.4 (2.1)

2. Primary Outcome: Change in Systolic Blood Pressure From Baseline to 4 Hours
Description: Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 8 hour infusion with subjects in supine position. Change is the difference between 4 hour systolic blood pressure from baseline systolic blood pressure.
Time Frame: Baseline, 4 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mmHg
  Saline | 1.92 (4.01)
  Intralipid 20% | 12.58 (2.1)
  Dextrose 10% | 3.00 (3.35)
  Intralipid/Dextrose | 1.91 (5.00)

3. Primary Outcome: Change in Systolic Blood Pressure From Baseline to 8 Hours
Description: Systolic blood pressure is the amount of pressure your heart generates when pumping blood through your arteries to the rest of your body. Current guidelines identify normal systolic blood pressure as lower than 120 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 8 hour infusion with subjects in supine position. Change is the difference between 8 hour systolic blood pressure from baseline systolic blood pressure.
Time Frame: Baseline, 8 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mmHg
  Saline | 0.33 (4.89)
  Intralipid 20% | 12.08 (2.48)
  Dextrose 10% | 2.58 (3.09)
  Intralipid/Dextrose | 12.9 (6.62)

4. Secondary Outcome: Change in FFA (Free Fatty Acid) Levels From Baseline to 4 Hours
Description: Blood samples were collected for measurement of free fatty acids (FFA) at baseline and 4 hours after each infusion. FFA levels were determined by colorimetric method. Current guidelines identify normal range of FFA level as less than 0.72 mmol/L. Elevated plasma levels of FFA indicate a greater rate of insulin resistance. Change is the difference between 4 hour FFA levels from baseline FFA levels.
Time Frame: Baseline, 4 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mmol/L
  Saline | -0.05 (0.27)
  Intralipid 20% | 0.84 (0.8)
  Dextrose 10% | -0.13 (0.43)
  Intralipid/Dextrose | -0.11 (0.48)

5. Secondary Outcome: Changes in FFA (Free Fatty Acid) Levels From Baseline to 8 Hours
Description: Blood samples were collected for measurement of free fatty acids (FFA) at baseline and 8 hours after each infusion. FFA levels were determined by colorimetric method. Current guidelines identify normal range of FFA level as less than 0.72 mmol/L. Elevated plasma levels of FFA indicate a greater rate of insulin resistance. Change iis the difference between 8 hour FFA levels from baseline FFA levels.
Time Frame: Baseline, 8 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mmol/L
  Saline | 0.03 (0.46)
  Intralipid 20% | 1.03 (1.1)
  Dextrose 10% | -0.18 (0.46)
  Intralipid/Dextrose | -0.1 (0.3)

6. Secondary Outcome: Change in Triglyceride Levels From Baseline to 4 Hours
Description: Blood samples were collected for measurement of triglycerides at baseline and 4 hours after each infusion. Triglyceride levels were measured on CX7 Chemistry Analyzer. Current guidelines identify normal range of triglyceride level as less than 150 mg/dL. Elevated levels of triglycerides are associated with an increased risk of developing heart disease. Change is the difference between 4 hour triglyceride levels from baseline triglyceride levels.
Time Frame: Baseline, 4 hours
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mg/dL
  Saline | -0.83 (37.7)
  Intralipid 20% | 118.9 (86.7)
  Dextrose 10% | -4.99 (51.2)
  Intralipid/Dextrose | 39.6 (30.56)

7. Secondary Outcome: Change in Triglyceride Levels From Baseline to 8 Hours
Description: Blood samples were collected for measurement of triglycerides at baseline and 4 hours after each infusion. Triglyceride levels were measured on CX7 Chemistry Analyzer. Current guidelines identify normal range of triglyceride level as less than 150 mg/dL. Elevated levels of triglycerides are associated with an increased risk of developing heart disease. Change is the difference between 8 hour triglyceride levels from baseline triglyceride levels.
Time Frame: Baseline, 8 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mg/dL
  Saline | 2.1 (38.3)
  Intralipid 20% | 121.1 (96.8)
  Dextrose 10% | 3.98 (62.3)
  Intralipid/Dextrose | 47.3 (50.7)

8. Secondary Outcome: Plasma Glucose Levels for Saline Infusion
Description: Blood samples were collected for measurement of plasma glucose levels at baseline, 4 hours after saline infusion, and 8 hours after saline infusion. Plasma glucose was measured on CX7 Chemistry Analyzer. Current guidelines identify normal fasting glucose as less than 100 mg/dL. High levels of glucose most frequently indicates diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mg/dL
  Baseline | 86.0 (9.6)
  4 hours | 87.0 (20.7)
  8 hours | 88.0 (15.0)

9. Secondary Outcome: Plasma Glucose Levels for Intralipid Infusion
Description: Blood samples were collected for measurement of plasma glucose levels at baseline, 4 hours after intralipid infusion, and 8 hours after intralipid infusion. Plasma glucose was measured on CX7 Chemistry Analyzer. Current guidelines identify normal fasting glucose as less than 100 mg/dL. High levels of glucose most frequently indicates diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mg/dL
  Baseline | 78.4 (8.0)
  4 hours | 75.6 (9.4)
  8 hours | 73.7 (10.6)

10. Primary Outcome: Change in Diastolic Blood Pressure From Baseline to 4 Hours
Description: Diastolic blood pressure is the amount of pressure in your arteries when your heart is at rest between beats. Current guidelines identify normal diastolic blood pressure as lower than 80 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 8 hour infusion with subjects in supine position. Change is the difference between 4 hour diastolic blood pressure from baseline diastolic blood pressure.
Time Frame: Baseline, 4 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mmHg
  Saline | -1.25 (2.7)
  Intralipid 20% | 6.2 (2.35)
  Dextrose 10% | -2.08 (9.26)
  Intralipid/Dextrose | -4.27 (14.95)

11. Primary Outcome: Change in Diastolic Blood Pressure From Baseline to 8 Hours
Description: Diastolic blood pressure is the amount of pressure in your arteries when your heart is at rest between beats. Current guidelines identify normal diastolic blood pressure as lower than 80 mmHg. Blood pressure was measured in triplicate with a manual cuff prior to and every 4 hours during the 8 hour infusion with subjects in supine position. Change is the difference between 8 hour diastolic blood pressure from baseline diastolic blood pressure.
Time Frame: Baseline, 8 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mmHg
  Saline | 1.2 (10.5)
  Intralipid 20% | 4.8 (6.2)
  Dextrose 10% | -0.83 (9.7)
  Intralipid/Dextrose | 2.7 (9.0)

12. Secondary Outcome: Plasma Glucose Levels for Dextrose Infusion
Description: Blood samples were collected for measurement of plasma glucose levels at baseline, 4 hours after dextrose infusion, and 8 hours after dextrose infusion. Plasma glucose was measured on CX7 Chemistry Analyzer. Current guidelines identify normal fasting glucose as less than 100 mg/dL. High levels of glucose most frequently indicates diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mg/dL
  Baseline | 77.4 (12.4)
  4 hours | 100.4 (19.5)
  8 hours | 93.0 (13.9)

13. Secondary Outcome: Plasma Glucose Levels for Intralipid/Dextrose Infusion
Description: Blood samples were collected for measurement of plasma glucose levels at baseline, 4 hours after intralipid/dextrose infusion, and 8 hours after intralipid/dextrose infusion. Plasma glucose was measured on CX7 Chemistry Analyzer. Current guidelines identify normal fasting glucose as less than 100 mg/dL. High levels of glucose most frequently indicates diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
mg/dL
  Baseline | 71.6 (12.3)
  4 hours | 101.2 (16.6)
  8 hours | 97.8 (11.1)

14. Secondary Outcome: Insulin Levels for Saline Infusion
Description: Blood samples were collected for the measurement of insulin levels at baseline, 4 hours after saline infusion, and 8 hours after saline infusion. Insulin was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal insulin levels as 8.8 μU/mL for men and 8.4 for women. High levels of insulin most frequently indicate insulin resistance or hypoglycemia, if paired with a low glucose level. Low levels of insulin paired with high glucose level can indicate diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
μU/mL
  Baseline | 8.4 (4.9)
  4 hours | 11.3 (6.4)
  8 hours | 10.1 (6.6)

15. Secondary Outcome: Insulin Levels for Intralipid Infusion
Description: Blood samples were collected for the measurement of insulin levels at baseline, 4 hours after intralipid infusion, and 8 hours after intralipid infusion. Insulin was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal insulin levels as 8.8 μU/mL for men and 8.4 for women. High levels of insulin most frequently indicate insulin resistance or hypoglycemia, if paired with a low glucose level. Low levels of insulin paired with high glucose level can indicate diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
μU/mL
  Baseline | 9.1 (5.5)
  4 hours | 11.3 (7.7)
  8 hours | 9.3 (7.5)

16. Secondary Outcome: Insulin Levels for Dextrose Infusion
Description: Blood samples were collected for the measurement of insulin levels at baseline, 4 hours after dextrose infusion, and 8 hours after dextrose infusion. Insulin was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal insulin levels as 8.8 μU/mL for men and 8.4 for women. High levels of insulin most frequently indicate insulin resistance or hypoglycemia, if paired with a low glucose level. Low levels of insulin paired with high glucose level can indicate diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
μU/mL
  Baseline | 8.4 (9.6)
  4 hours | 25.1 (10.2)
  8 hours | 33.4 (21.0)

17. Secondary Outcome: Insulin Levels for Intralipid/Dextrose Infusion
Description: Blood samples were collected for the measurement of insulin levels at baseline, 4 hours after intralipid/dextrose infusion, and 8 hours after intralipid/dextrose infusion. Insulin was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal insulin levels as 8.8 μU/mL for men and 8.4 for women. High levels of insulin most frequently indicate insulin resistance or hypoglycemia, if paired with a low glucose level. Low levels of insulin paired with high glucose level can indicate diabetes.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
μU/mL
  Baseline | 10.4 (9.6)
  4 hours | 28.0 (12.5)
  8 hours | 40.5 (22.8)

18. Secondary Outcome: C-peptides Levels for Saline Infusion
Description: Blood samples were collected for the measurement of C-peptide levels at baseline, 4 hours after saline infusion, and 8 hours after saline infusion. C-peptide was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal C-peptide levels as 0.51 to 2.72 ng/mL.
  A high level of C-peptide generally indicates a high level of endogenous insulin production. This may be in response to a high blood glucose caused by glucose intake and/or insulin resistance. A high level of C-peptide is also seen with insulinomas and may be seen with low blood potassium, Cushing syndrome, and renal failure. A low level of C-peptide is associated with a low level of insulin production. This can occur when insufficient insulin is being produced by the beta cells, with diabetes for example, or when production is suppressed by treatment with exogenous insulin.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
ng/mL
  Baseline | 2.21 (1.04)
  4 hours | 2.06 (0.96)
  8 hours | 2.71 (1.36)

19. Secondary Outcome: C-peptides Levels for Intralipid Infusion
Description: Blood samples were collected for the measurement of C-peptide levels at baseline, 4 hours after Intralipid infusion, and 8 hours after Intralipid infusion. C-peptide was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal C-peptide levels as 0.51 to 2.72 ng/mL.
  A high level of C-peptide generally indicates a high level of endogenous insulin production. This may be in response to a high blood glucose caused by glucose intake and/or insulin resistance. A high level of C-peptide is also seen with insulinomas and may be seen with low blood potassium, Cushing syndrome, and renal failure. A low level of C-peptide is associated with a low level of insulin production. This can occur when insufficient insulin is being produced by the beta cells, with diabetes for example, or when production is suppressed by treatment with exogenous insulin.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
ng/mL
  Baseline | 2.14 (1.12)
  4 hours | 2.39 (1.16)
  8 hours | 2.40 (1.23)

20. Secondary Outcome: C-peptides Levels for Dextrose Infusion
Description: Blood samples were collected for the measurement of C-peptide levels at baseline, 4 hours after dextrose infusion, and 8 hours after dextrose infusion. C-peptide was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal C-peptide levels as 0.51 to 2.72 ng/mL.
  A high level of C-peptide generally indicates a high level of endogenous insulin production. This may be in response to a high blood glucose caused by glucose intake and/or insulin resistance. A high level of C-peptide is also seen with insulinomas and may be seen with low blood potassium, Cushing syndrome, and renal failure. A low level of C-peptide is associated with a low level of insulin production. This can occur when insufficient insulin is being produced by the beta cells, with diabetes for example, or when production is suppressed by treatment with exogenous insulin.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
ng/mL
  Baseline | 1.96 (1.58)
  4 hours | 4.73 (1.61)
  8 hours | 5.79 (2.08)

21. Secondary Outcome: C-peptides Levels for Intralipid/Dextrose Infusion
Description: Blood samples were collected for the measurement of C-peptide levels at baseline, 4 hours after intralipid/dextrose infusion, and 8 hours after intralipid/dextrose infusion. C-peptide was measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the DPC Immulite analyzer. Current guidelines identify normal C-peptide levels as 0.51 to 2.72 ng/mL.
  A high level of C-peptide generally indicates a high level of endogenous insulin production. This may be in response to a high blood glucose caused by glucose intake and/or insulin resistance. A high level of C-peptide is also seen with insulinomas and may be seen with low blood potassium, Cushing syndrome, and renal failure. A low level of C-peptide is associated with a low level of insulin production. This can occur when insufficient insulin is being produced by the beta cells, with diabetes for example, or when production is suppressed by treatment with exogenous insulin.
Time Frame: Baseline, 4 hours, 8 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 12
ng/mL
  Baseline | 2.23 (1.52)
  4 hours | 4.97 (1.74)
  8 hours | 6.43 (2.41)

ADVERSE EVENTS:
Arm/Group | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
A larger sample size and inclusion of subjects from different ethnicities would be required to generalize the results of this study. Study used healthy volunteers--outcomes cannot be applied to patients with diabetes mellitus or insulin resistance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes